CLINICAL TRIAL: NCT06297265
Title: Feasibility and Effects of Manual Lymphatic Drainage (MLD) Breast Massage in Breast Cancer Patients Undergoing Adjuvant Radiation Therapy
Brief Title: Manual Lymphatic Drainage Breast Massage in Breast Cancer Patients After Breast Conserving Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-23-2; NCI-2023-10828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-23-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2024-02-09; First posted 2024-03-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Localized Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Supportive care (MLD breast massage) (Experimental): Patients undergo MLD breast massage over 30-60 minutes BIW for the duration of SOC radiation therapy and for 1 month thereafter.
  Interventions: Other: Lymphedema Management; Other: Questionnaire Administration; Radiation: Adjuvant breast radiation therapy

INTERVENTIONS:
Other: Lymphedema Management — Undergo MLD breast massage
Other: Questionnaire Administration — Ancillary studies
Radiation: Adjuvant breast radiation therapy — Using standard 3D conformal or intensity modulated techniques, patients will receive standard fractionation or moderate hypofractionation radiation therapy. The radiation treatment will last for 3 to 6 weeks, with the length of treatment depending on patient's specific clinical situation.
  Other Names: Radiotherapy

SUMMARY:
This phase II trial evaluates manual lymphatic drainage breast massage for reducing treatment-related side effects in women undergoing radiation therapy after breast conserving surgery for breast cancer that has not spread to other parts of the body (localized). Breast conserving surgery can be an effective treatment option for early stage breast cancer, but it can also be associated with side effects including fluid collection in tissues/swelling (lymphedema), pain, reduced quality of life, and poorer body image. Manual lymphatic drainage is a gentle massage technique used to reduce swelling. It may be a safe and effective way to reduce treatment-related side effects in women receiving radiation therapy after surgery for localized breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of breast manual lymphatic drainage (MLD) on breast cancer patients receiving adjuvant breast radiation therapy after breast conserving surgery.

SECONDARY OBJECTIVES:

I. Evaluate the tolerability of breast manual lymphatic drainage (MLD) on breast cancer patients receiving adjuvant breast radiation therapy after breast conserving surgery.

II. Preliminarily assess the effect on acute and chronic breast edema, pain, functional status, quality of life, body image and radiation induced fibrosis (RIF).

OUTLINE:

Patients undergo MLD breast massage over 30-60 minutes twice a week (BIW) for the duration of standard of care (SOC) radiation therapy and for 1 month thereafter.

After completion of SOC radiation therapy, patients are followed up at 2-4 weeks and 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female with native breasts and localized breast cancer who are status post-lumpectomy surgery, will receive whole breast radiation therapy with/without nodal irradiation, with standard fractionation or moderate hypofractionation
* Age >= 18 years
* Ability to understand and the willingness to sign a written informed consent in English or Spanish

Exclusion Criteria:

* Underlying diagnosis of chronic inflammatory illness or collagen vascular disorder, e.g. scleroderma, lupus, rheumatoid arthritis, fibromyalgia as these conditions may significantly affect the likelihood and magnitude of radiation related toxicity
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Inability to provide written informed consent in English or Spanish
* Patients receiving ultra-hypofractionation, and/or partial breast or chest wall radiation therapy are excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be female with native breasts. Cis males, transgender females, and cis females without intact native breasts are excluded.
Enrollment: 50 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2027-05-24 (Estimated)

PRIMARY OUTCOMES:
Rate of compliance of MLD breast massage sessions | Up to 1 month after completion of radiation
  The intervention compliance rate will be calculated as the percentage of completed treatment sessions over the total targeted treatment sessions.

SECONDARY OUTCOMES:
Assess the effect of MLD breast massage breast edema | Up to 1 year
  The Dutch Breast Edema Questionnaire (BrEQ-Dutch version) will be used to diagnose the presence of breast edema. Getting 8.5 points from the questionnaire is the cut-off point. There is no breast edema below 8.5, there is breast edema above 8.5. It has a score between 0-80 points. Higher total symptom score means worse edema.
Assess the effect of MLD breast massage on pain | Up to 1 year
  Pain will be graded using NCI-CTCAE version 5.0
Assess the effect of MLD breast massage on functional status | From baseline to follow-up (2-4 weeks, and 3, 6, and 12 months)
  Will be assessed using the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire. The FACT-B consists of 37 questions that address physical, social, emotional, and functional well-being. Each item has a score range of 0 (Not at all) to 4 (Very much), with a total score ranging from 0-148 The higher the score, the better the QOL reported by the participant.
Assess the effect of MLD breast massage on quality of life | From baseline to follow-up (2-4 weeks, and 3, 6, and 12 months)
  Quality of Life will be assessed using the European Quality of Life 5 Dimension 5 Level (EuroQoL EQ-5D-5L) questionnaire. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems (1-5). The patient is asked to indicate her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A higher score indicates more severe or frequent problems.
Assess the effect of MLD breast massage on body image | From baseline to follow-up (2-4 weeks, and 3, 6, and 12 months)
  Will be assessed using the Body Image Scale (BIS). The 10-item Body Image Scale was developed by Hopwood et al. in 2001 to measure affective, behavioral, and cognitive body image symptoms. Patients can indicate body image symptoms on a 4-point scale (0 "not at all" to 3 "very much"). The total score ranges from 0 to 30 and can be calculated by summing up the 10 items. A higher score means a higher level of body image disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: May L Tao, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States